CLINICAL TRIAL: NCT02794675
Title: A Pilot Study Using Intraoperative Placement of Cesium-131 Permanent Interstitial Brachytherapy in Resectable High Risk Recurrent Head and Neck Cancer
Brief Title: Intraoperative Placement of Cesium-131 Permanent Interstitial Brachytherapy in Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5315; NCI-2017-00023 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: resectable; Cesium 131; brachytherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cesium-131; Cesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cesium 131 brachytherapy (Experimental): Cesium 131 is the radioactive isotope in the protocol. The prescribed dose will range from 50-80 Gy at maximal delivery. It comes in 0.5 cm seeds that will be placed in the tumor resection bed at 1cm intervals. They are implantable seeds that do not require removal.
  Interventions: Drug: Cesium 131

INTERVENTIONS:
Drug: Cesium 131 — The number sources and activity will be based on the target volume to deliver total radiation dose, this will vary per patient.
  Other Names: Cs-131; Cesium

SUMMARY:
The purpose of this study is to explore the use of a treatment called interstitial brachytherapy for patients who have a high risk resectable (able to be treated with surgery) recurrent head and neck cancer.

Brachytherapy is a form of radiation therapy that uses radioactive seeds and implants them into a specific place on your body. This study is using Cesium-131 permanent interstitial brachytherapy.

Cesium-131 is FDA approve for brachytherapy use, however, there are currently no research studies to show how effective it is for head and neck cancer. The goal of this study is determine the effect that the placement of Cesium-131 brachytherapy seeds has on overall survival as well as to assess possible side effects.

DETAILED DESCRIPTION:
Primary Objective:

To assess the effect of Cesium 131 brachytherapy in subjects with resectable recurrent cancer of the head and neck by evaluating disease free survival (DFS) and comparing to a previous cohort. Potential effects on locoregional control rate and overall survival will be explored.

Secondary Objective:

To assess toxicity associated with cesium 131 brachytherapy treatment.

Study Design Patients with a head and neck recurrent cancer who are planned to undergo definitive tumor resection surgery that meet our inclusion and exclusion criteria will be offered participation in this clinical trial.

Participant's Follow-up. The participant's medical records will be reviewed every 3 months for 24 months to assess: loco-regional control, distant metastasis free survival, disease free survival, and overall survival. This will allow us to assess the potential treatment effect of cesium 131.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed recurrent head and neck cancer.
* Based on clinical and radiographic evidence the tumor needs to be deemed resectable preoperatively by the surgeon and when necessary (determined by the surgeon) tumor board review.
* Patients must have potentially curable disease
* Karnofsky Performance status ≥ 60% (ECOG/Zubrod 0,1,or 2)
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 7.0 g/dl
  * Absolute neutrophil count (ANC) > 500/mcL
  * Platelet count ≥ 75,000/mcL
* Patients with recurrent/previous treated head and neck squamous cell carcinoma that is deemed surgically resectable by the treating physician but at high risk for recurrence due to concerns regarding close and/or margins due to locations on or near critical structures such as internal or common carotid, skull base, deep cervical musculature, and other areas that may limit the possibility of an enbloc resection. This group otherwise would be considered for retreatment with radiation and/or chemoradiation.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients deemed to have un-resectable disease by the treating surgeon or upon tumor board review.

  * Patients with exposed carotid artery preoperatively requiring sacrifice or bypass intra-operatively
  * Patients with active pharyngocutaneous fistula
  * Patients may have had a recent previous hospital admission (within 30 days) or be admitted preoperatively but not for the following conditions

    * Unstable angina
    * Congestive heart failure
    * Severe hypothyroidism TSH >10

      ---- Endocrine consult and intervention may allow participation at the discretion of the principal investigator for a thyroid-stimulating hormone (TSH) > 10.
    * Patients deemed to be "High Risk" by pre admission testing (CPM) or by a preoperative risk assessment by the hospitalist for perioperative complications
    * Subjects with more than one site of distant metastatic disease (beyond the head and neck) as evidenced by computerized tomography (CT) scan or positron emission tomography/CT (PET/CT) or biopsy ---- A subject with a single lung nodule (deemed cancerous by PET/CT or Biopsy) will not be excluded.
* Subjects receiving any other investigational agents.
* Subjects with untreated brain metastases/central nervous system disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cesium 131 or other agents used in this study.
* Pregnant or breastfeeding women are excluded from this study because Cesium 131 has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with Cesium 131, breastfeeding should be discontinued if the mother is treated with Cesium 131. These potential risks may also apply to other agents used in this study.
* Subjects who are HIV-positive will be excluded from the study. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Cesium 131. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Median disease free survival (DFS) | Up to two years
  DFS defined as the time of diagnosis with no evidence of disease through death by any cause or relapse of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Min Yao, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Luginbuhl A, Calder A, Kutler D, Zender C, Wise-Draper T, Patel J, Cheng M, Karivedu V, Zhan T, Parashar B, Gulati S, Yao M, Lavertu P, Takiar V, Tang A, Johnson J, Keane W, Curry J, Cognetti D, Bar-Ad V. Multi-Institutional Study Validates Safety of Intraoperative Cesium-131 Brachytherapy for Treatment of Recurrent Head and Neck Cancer. Front Oncol. 2021 Nov 26;11:786216. doi: 10.3389/fonc.2021.786216. eCollection 2021. PMID 34900741
- [Derived] Kharouta M, Zender C, Podder T, Rezaee R, Lavertu P, Fowler N, Thuener J, Li S, Clancy K, Xu Z, Yao M. Permanent Interstitial Cesium-131 Brachytherapy in Treating High-Risk Recurrent Head and Neck Cancer: A Prospective Pilot Study. Front Oncol. 2021 Mar 18;11:639480. doi: 10.3389/fonc.2021.639480. eCollection 2021. PMID 33816283